CLINICAL TRIAL: NCT03635892
Title: A Phase 2 Open-Label Study of Nivolumab Combined With Cabozantinib in Subjects With Advanced or Metastatic Non-Clear Cell Renal Cell Carcinoma (CA209-9KU)
Brief Title: A Study of Nivolumab In Combination With Cabozantinib in Patients With Non-Clear Cell Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-254
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Advanced or Metastatic Non-clear Cell Renal Cell Carcinoma; Unclassified Renal Cell Carcinoma; Papillary Renal Cell Carcinoma; Fumarate Hydratase Deficient Renal Cell Carcinoma; Succinate Dehydrogenase Deficient Renal Cell Carcinoma; Collecting Duct Renal Cell Carcinoma; Chromophobe Renal Cell Carcinoma
Keywords: Nivolumab; Cabozantinib; 18-254
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a single institution open-label phase II trial of cabozantinib and nivolumab in patients with advanced or metastatic non-clear cell Renal Cell Carcinoma (nccRCC), who have not received prior PD-1/PD-L1 directed therapy. This study is designed as separate cohorts defined by histology across three cohorts.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Unclassified, papillary, and HL RCC (Experimental): Cohort 1 is designed as a single stage study with a total sample size of 20. This design discriminates between ORR rates of 10 and 35%.
  Interventions: Drug: cabozantinib; Drug: nivolumab
- Cohort 2: Chromophobe RCC (Experimental): Cohort 2 is designed as a Simon's optimal two-stage design with a total possible sample size of 17. This design discriminates between ORR rates of 5 and 25%.
  Interventions: Drug: cabozantinib; Drug: nivolumab
- Cohort 3: Unclassified, papillary, and HL RCC (Experimental): Cohort 3 is designed as an expansion cohort of Cohort 1 with 20 additional patients to obtain a more precise estimate of the ORR and clinical outcomes
  Interventions: Drug: cabozantinib; Drug: nivolumab
- Cohort 4: Unclassified, papillary, and HL RCC (Experimental): Cohort 4 is an expansion of Cohorts 1+3, which will accure an additional 40 patients
  Interventions: Drug: cabozantinib; Drug: nivolumab

INTERVENTIONS:
Drug: cabozantinib — cabozantinib 40mg, self administered orally once daily on a continuous schedule (days 1-28) Patients will continue to take cabozantinib until disease progression (unless continuing treatment beyond progression), major toxicity, or withdrawal from the study for any reason.
  Other Names: CABOMETYX®
Drug: nivolumab — Patients will receive an intravenous infusion of nivolumab, per institutional standards, at 240 mg on Cycle 1, Day 1 and will return to the center approximately every two weeks (14 ± 3 days) for subsequent infusions until disease progression (unless continuing treatment beyond progression), major toxicity, or withdrawal from the study for any reason.
  Other Names: Opdivo

SUMMARY:
The purpose of this study is to compare any good and bad effects of using a combination of nivolumab (Opdivo®) and cabozantinib (Cabometyx®) in people with metastatic kidney cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated IRB-approved Informed Consent Form
* Pathologic or histologically confirmed unresectable advanced or metastatic nccRCC
* 0 or 1 prior systemic therapies, including treatment in the adjuvant setting
* Availability of a representative formalin fixed, paraffin embedded tumor specimen or fresh frozen tissue specimen that enables the definitive diagnosis of RCC, accompanied by an associated pathology report. Specimens can be collected by surgical resection or biopsy of the primary tumor or biopsy or resection of a metastatic lesion.
* Measurable disease, as defined by RECIST 1.1
* Age ≥18 years
* KPS ≥ 70
* Recovery to baseline or ≤ Grade 1 CTCAE v4 from toxicities related to any prior treatments, unless adverse events (AE(s)) are clinically nonsignificant and/or stable on supportive therapy.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:

  * ANC ≥ 1500 cells/μL (without granulocyte colony stimulating factor support within 2 weeks prior to Cycle 1, Day 1)
  * WBC counts ≥ 2500/μL and ≤ 15,000/μL without G-CSF
  * Lymphocyte count ≥ 500/μL
  * Platelet count ≥100,000/μL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
  * Hemoglobin ≥9.0 g/dL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN). ALP ≤ 5 x ULN if patient has documented bone metastases.
* Serum bilirubin ≤ 1.5 x ULN . Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
* Serum albumin ≥ 2.8 g/dl
* Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
* INR and aPTT ≤ 1.3 x ULN • within 14 days of first dose of study treatment.This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
* Creatinine ≤ 2.0 x ULN or Calculated Creatinine clearance ≥ 30mL/min
* For women who are not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use two adequate methods of contraception, including at least one method with a failure rate of ≥ 1% per year
* Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol)
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 5 months after the last dose of study treatment for females and 7 months for males.
* Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who are surgically sterile as described above).

However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.

* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.

Exclusion Criteria:

* Prior treatment with an immunotherapy agent including high dose IL-2, anti-CTLA-4, anti-PD1, and anti-PD-L1 agents
* Prior treatment with cabozantinib for non-clear cell RCC
* Receipt of any type of small molecule kinase inhibitor within 2 weeks of treatment.
* Receipt of any type of anti-cancer antibody, cytotoxic anticancer therapy, or any other investigational agents within 4 weeks of treatment start
* Known malignancies of the brain or spinal cord or leptomeningeal disease
* Patients requiring pain medication must be on a stable regimen at study entry
* Systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroids > 10 mg daily prednisone equivalents are allowed in the absence of autoimmune disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled hypercalcemia (≥ 1.5 mmol/L ionized calcium or Ca ≥ 12 mg/dL or corrected serum calcium ≥ ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
* Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy
* Pregnant and lactating women History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of HIV infection
* Patients with active or chronic hepatitis B or hepatitis C infection
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 6 months, unstable arrhythmias, unstable angina, or EF < 50%
* Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment
* Patients with known coronary artery disease, congestive heart failure not meeting the above criteria must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
* Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (eg, simple excision, biopsy, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* History of stroke or transient ischemic attack within 6 months prior to Cycle 1, Day 1
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Patients with a history of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to study enrollment
* Other clinically significant disorders that would preclude safe study participation

  * Serious non-healing wound/ulcer/bone fracture
  * Uncompensated/symptomatic hypothyroidism
  * Moderate to severe hepatic impairment (Child-Pugh B or C)
* Corrected QT interval calculated by the Frederica formula (QTcF) > 500 ms per elFectrocardiogram (ECG) within 28 days before first dose of study treatment Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility
* Inability to swallow tablets or capsules
* Previously identified allergy or hypersensitivity to components of the study treatment formulations
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Low-dose aspirin for cardio protection (per local applicable guidelines) is permitted
  * Low-dose low molecular weight heparins (LMWH) are permitted
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 1 week before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
* The subject has tumor invading or encasing any major blood vessels
* The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* Uncontrolled hypertension (>150 mmHg systolic or > 100 mmHg diastolic despite optimal antihypertensive treatment)
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible. Radiation for palliation is allowable on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 2 years
  per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Lee CH, Voss MH, Carlo MI, Chen YB, Zucker M, Knezevic A, Lefkowitz RA, Shapnik N, Dadoun C, Reznik E, Shah NJ, Owens CN, McHugh DJ, Aggen DH, Laccetti AL, Kotecha R, Feldman DR, Motzer RJ. Phase II Trial of Cabozantinib Plus Nivolumab in Patients With Non-Clear-Cell Renal Cell Carcinoma and Genomic Correlates. J Clin Oncol. 2022 Jul 20;40(21):2333-2341. doi: 10.1200/JCO.21.01944. Epub 2022 Mar 17. PMID 35298296
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm